CLINICAL TRIAL: NCT05540392
Title: Nocturia in Prostate Cancer Survivors - Acupuncture Pilot Study (NOCTURNAL)
Brief Title: An Acupuncture Study for Prostate Cancer Survivors With Urinary Issues
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-270
Record Dates: First submitted 2022-09-09; First posted 2022-09-14 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Survivorship; Prostate Cancer
Keywords: Acupuncture; Urinary issue; Nocturia; 22-270
MeSH Terms: conditions — Prostatic Neoplasms; Nocturia | interventions — Acupuncture Therapy; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): Acupuncture group will receive 10 treatments of acupuncture over the course of 10 weeks (i.e. one treatment a week) with a +/- 14-day window.
  Interventions: Procedure: Acupuncture; Other: Questionnaires
- Waitlist Control (Experimental): The waitlist control group will not receive any acupuncture treatments during the 14-week waiting period. Patients in waitlist control group will have the option to receive up to 10 acupuncture treatments after a 14-week waiting period.
  Interventions: Other: Waitlist Control; Other: Questionnaires

INTERVENTIONS:
Procedure: Acupuncture — 10 treatments of acupuncture over the course of 10 weeks
  Arms: Acupuncture
Other: Waitlist Control — The waitlist control group will not receive any acupuncture treatments during the 14-week waiting period. Patients in waitlist control group will have the option to receive up to 10 acupuncture treatments after a 14-week waiting period.
  Arms: Waitlist Control
Other: Questionnaires — Patients will complete Patient Reported Outcomes (PRO)

SUMMARY:
The purpose of this study is to test whether acupuncture can improve nocturia in prostate cancer survivors. This is the first time acupuncture is being studied for nocturia in prostate cancer survivors. Researchers will see if acupuncture is a practical treatment option for prostate cancer survivors with nocturia. The study will also look at the effect acupuncture has on nocturia and other symptoms prostate cancer survivors experience such as insomnia, hot flashes, anxiety, depression, tiredness (fatigue), sexual dysfunction, and cognitive (mental) difficulties.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Prior PC diagnosis
* No evidence of Prostate Cancer
* Clinically meaningful nocturia, defined as ≥2 nocturia episodes every night for the past month

Exclusion Criteria:

* <1 month since completion of PC treatment (surgery, chemotherapy, radiation, ADT)
* Score of ≥5 on the STOP-Bang questionnaire indicative of high risk of moderate-to severe obstructive sleep apnea
* Other untreated primary sleep disorder (e.g. delayed/advanced sleep phase syndrome)
* Untreated primary psychiatric disorder (e.g. bipolar disorder, schizophrenia, substance abuse, dementia)
* Initiation of new medications for urinary symptoms in the past 4 weeks
* Altered dosing of medications for urinary symptoms in the past 4 weeks
* Plan to initiate/change medications or other treatments (e.g. surgery, behavioral intervention, complementary therapies) for urinary symptoms during the study
* Implanted electronically charged medical device
* Unable to provide consent for himself
* Unwilling to adhere to all study-related procedures

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer
Enrollment: 60 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
success | 1 year
  If a participant completes at least 8 out of 10 acupuncture sessions. Feasibility will be evaluated based on the respective definitions of success for the acupuncture.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Liou, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center Suffolk - Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - MSK at Ralph Lauren (Consent Only), New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm